CLINICAL TRIAL: NCT03505216
Title: Swiss Paediatric Airway Cohort
Acronym: SPAC
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: SPAC
Record Dates: First submitted 2018-04-02; First posted 2018-04-23 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Asthma; Wheezing; Cough; Exercise Induced Bronchospasm; Inspiratory Laryngeal Obstruction; Dysfunctional Breathing
MeSH Terms: conditions — Asthma; Respiratory Sounds; Cough; Asthma, Exercise-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient population: Children referred to paediatric pulmonary outpatient clinics for respiratory symptoms such as wheeze, cough, dyspnea, exercise- and sleep-related breathing problems.

SUMMARY:
The Swiss Paediatric Airway Cohort (SPAC) is a national, prospective clinical cohort of children and adolescents who visit physicians in Switzerland for recurrent wheeze, cough, and exercise- or sleep-related respiratory problems. SPAC aims to answer important questions on clinical phenotypes, prognosis, diagnosis and treatment. SPAC is part of routine care, and only clinically indicated investigations are done. The comprehensive baseline assessment includes a detailed questionnaire to families, plus test results, diagnoses and treatments from hospital records. Follow-up is via monthly questionnaires the first 12 months and thereafter annual questionnaires to families, and data from follow-up visits.

Currently, 4344 patients from 10 clinics and hospitals in Switzerland (Aarau, Basel, Bern, Chur, Horgen, Lausanne, Luzern, St. Gallen, Worb, Zurich) have been enrolled.

SPAC provides real-life data on children visiting the Swiss health care system for common respiratory problems. It will provide a research platform for health services research, and for nested clinical and transitional studies.

Publications and plain language summaries are listed on the study website: https://www.spac-study.ch/publikationen/

DETAILED DESCRIPTION:
Background:

Many studies have investigated the epidemiology of asthma in childhood, but most were based on data from the general population gathered either in cross-sectional or longitudinal surveys in schoolchildren.

Objectives:

The Swiss Paediatric Airway Cohort (SPAC) was set up in 2017 as a large, longitudinal database that is representative of children and adolescents visiting physicians in Switzerland for recurrent wheeze, cough, and exercise- or sleep-related respiratory symptoms. It will constitute a national research platform for studying healthcare provision, phenotypes and prognosis of these problems, and a sampling frame for conducting nested studies.

Methods:

Recruitment and participation:

The SPAC study recruits patients aged 0-16 that are referred to a paediatric outpatient clinic for recurrent respiratory symptoms. Families receive a SPAC information package containing an invitation letter, study information leaflet, informed consent form, and questionnaire. Physicians introduce the study to them, answer questions, and collect informed consent forms. Completed questionnaires are brought by families to the clinics or sent directly by families to the SPAC study centre using a prepaid return envelope. Eligible patients have consultations in participating clinics regardless of their study participation. No tests are performed specifically for SPAC; examinations and tests are done only if clinically indicated or ordered by the referring physician. Examinations such as lung function, allergy, blood, or bronchial challenge tests are done using respective standard procedures in the clinics. SPAC research team members visit participating centres at regular intervals to collect data. During the first year, caregivers or patients who are 14 years or older receive short online questionnaire through a link via email. One year after enrolment and each year thereafter, caregivers receive a follow-up questionnaire by post.

Information collected:

Questionnaires:

At baseline families complete a detailed questionnaire that includes sections on frequency, duration, severity, triggers, and history of upper and lower respiratory symptoms, and diagnoses, treatments, health behaviours, environmental factors, family history, and contact information. The monthly online questionnaires focus on symptoms, infections, and treatments which may change short-term. The yearly follow-up questionnaires focus on symptoms, treatments, and important risk factors during the past 12 months. Postal addresses for mailing are obtained from hospital records and updated by contacting community registration offices, a procedure used successfully for other registries and cohort studies in Switzerland. Questionnaires are currently available in German and French.

Medical records:

Information obtained from medical records includes reasons for referral; anthropometric measures; results from the physical examination and diagnostic tests including pulmonary function, allergy, and blood tests; information about asthma control; and final diagnoses and prescribed treatments.

Linkage to routine data:

For specific analyses, probabilistic record linkage will be used to merge data from SPAC with routine datasets collected by the Swiss Federal Statistical Office.

Study database:

The SPAC database is web-based, using the Research Electronic Data Capture (REDCap) platform developed at Vanderbilt University. REDCap is widely used in academic research and allows data entry and extraction in various formats.

Current status of the project:

SPAC recruits participants from 10 clinics in Switzerland including the children's hospital in Aarau, the University Children's hospital in Basel, the University Children's Hospital in Bern, the Children's hospital in Chur, a private paediatric pulmonology clinic in Horgen, the University Children's hospital in Lausanne, the Children's hospital in Luzern, the Children's hospital in St. Gallen, a private paediatric pulmonology clinic in Worb, and the University Children's Hospital in Zurich. By October 2023, 4344 children have agreed to participate in SPAC.

Publications and plain language summaries are listed on the study website: https://www.spac-study.ch/publikationen/

Funding:

Setting up SPAC was funded by the Swiss National Science Foundation (SNF32003B_162820, SNF320030_182628, SNF320030_212519), and several local funding bodies including the Swiss Lung Association, the Lung League of St. Gallen, and the Allergiestiftung Ulrich Müller-Gierok.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 0-16 years
* Resident in Switzerland
* Seen in a paediatric pulmonary outpatient clinic due to respiratory problems
* Parents and patients above age 14 must be able to sign an informed consent form

Exclusion Criteria:

Prior diagnosis of cystic fibrosis, primary ciliary dyskinesia, severe heart disease, oncological disease, neuromuscular disease or severe disability

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric pulmonology outpatient clinics in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2017-06-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Wheeze | 1 year from inclusion in SPAC study
  Number of patients with current wheeze as measured with questionnaire
Cough apart from colds | 1 year from inclusion in SPAC study
  Number of patients with cough apart from colds as measured with questionnaires
Exercise-induced dyspnea | 1 year from inclusion in SPAC study
  Number of patients with exercise-induced dyspnea as measured with questionnaires
Reduced lung function | 1 year from inclusion in SPAC study
  Number of patients with reduced lung function measured through clinical tests in the paediatric pulmonary clinics (Spirometry, Fraction of Exhaled Nitric Oxide, Bronchial challenge test, Exercise challenge test). Information collected through hospital records.

SECONDARY OUTCOMES:
Wheeze | 5 years from inclusion in SPAC study
  Number of patients with current wheeze as measured with questionnaire
Cough apart from colds | 5 years from inclusion in SPAC study
  Number of patients with Cough apart from colds as measured with questionnaire
Exercise-induced dyspnea | 5 years from inclusion in SPAC study
  Number of patients with Exercise-induced dyspnea as measured with questionnaire
Reduced lung function | 5 years from inclusion in SPAC study
  Number of patients with reduced lung function measured through clinical tests in the paediatric pulmonary clinics (Spirometry, Fraction of Exhaled Nitric Oxide,

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Kuehni, Prof., Study Director — Institute of Social and Preventive Medicine
Locations (12):
- Vienna Open Medical Institute, Vienna, Austria
- Switzerland (11):
  - Children's hospital Aarau, Aarau
  - University Children's hospital Basel, UKBB, Basel
  - Institute of Social and Preventive Medicine, Bern
  - University Children's Hospital Bern, Inselspital, Bern
  - Children's Hospital Chur, Chur
  - Pulmonology clinic, Horgen, Horgen
  - University Children's hospital Lausane, CHUV, Lausanne
  - Children's hospital Lucerne, Lucerne
  - Children's hospital St. Gallen, Sankt Gallen
  - Pulmonology clinic, Worb, Worb
  - University Children's Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Researchers who wish to develop a nested study with inclusion of additional data also need to submit a proposal to the SPAC committee and request permission. A concept sheet describing the planned analyses must be approved by the SPAC committee. If any additional data are collected by nested studies, these must be contributed to the SPAC database after the data collection. Nested studies might need separate ethics permission.
  At the study website: www.spac-study.ch, information can be found on how to request permission to use data from the SPAC study.

REFERENCES:
- See also: Study website — https://spac-study.ch/